CLINICAL TRIAL: NCT05877417
Title: The Chronic Effects of Low-Load Blood Flow Restriction and Creatine Supplementation in Women
Brief Title: Blood Flow Restriction and Creatine Supplementation in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, Paola Rivera, PhD Candidate, University of Central Florida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY00005471
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Physical Inactivity
Keywords: creatine; blood flow restriction; exercise
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Creatine; Blood Flow Restriction Therapy; Exercise

STUDY DESIGN:
Intervention Model Description: double blind placebo controlled
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (5):
- Control (No Intervention): If you are in the control group, there will be no supplement or exercise procedures.
  You will be asked to come in to the lab for 5 visits
- Creatine and Blood Flow Restriction Exercise (Experimental): * Of the other four groups, regardless of randomization, all 4 groups will be supplementing the same for the loading phase and throughout the study. Since this study is blinded, the research personnel will not know which supplement you are given and will therefore ensure everyone is following the same procedures.
  * Loading here means to consume more than the daily amount of supplement. This visit will have participants consume 5g twice in one day and twice more at home. This is a normal practice and standard use of the supplement.
  * If you are not in the control group, you will further be randomized into one of four possible supplementation groups. These groups will be double blinded and randomized into either placebo or creatine supplementation. Creatine monohydrate powder (Muscle Feast, Creapure®) will be used for the active supplement group. Dextrose powder (sugar) will be used for the placebo group.
  * The supplement and placebo are flavorless and odorless powder.
  Interventions: Dietary Supplement: Creatine Monohydrate; Device: Blood Flow Restriction
- Creatine and No-BFR with Training (Active Comparator): * Of the other four groups, regardless of randomization, all 4 groups will be supplementing the same for the loading phase and throughout the study. Since this study is blinded, the research personnel will not know which supplement you are given and will therefore ensure everyone is following the same procedures.
  * Loading here means to consume more than the daily amount of supplement. This visit will have participants consume 5g twice in one day and twice more at home. This is a normal practice and standard use of the supplement.
  * If you are not in the control group, you will further be randomized into one of four possible supplementation groups. These groups will be double blinded and randomized into either placebo or creatine supplementation. Creatine monohydrate powder (Muscle Feast, Creapure®) will be used for the active supplement group. Dextrose powder (sugar) will be used for the placebo group.
  * The supplement and placebo are flavorless and odorless powder.
  Interventions: Dietary Supplement: Creatine Monohydrate
- Placebo and Blood Flow Restriction Exercise (Placebo Comparator): * Of the other four groups, regardless of randomization, all 4 groups will be supplementing the same for the loading phase and throughout the study. Since this study is blinded, the research personnel will not know which supplement you are given and will therefore ensure everyone is following the same procedures.
  * Loading here means to consume more than the daily amount of supplement. This visit will have participants consume 5g twice in one day and twice more at home. This is a normal practice and standard use of the supplement.
  * If you are not in the control group, you will further be randomized into one of four possible supplementation groups. These groups will be double blinded and randomized into either placebo or creatine supplementation. Creatine monohydrate powder (Muscle Feast, Creapure®) will be used for the active supplement group. Dextrose powder (sugar) will be used for the placebo group.
  * The supplement and placebo are flavorless and odorless powder.
  Interventions: Device: Blood Flow Restriction
- Placebo and No-BFR with Training (Sham Comparator): * Of the other four groups, regardless of randomization, all 4 groups will be supplementing the same for the loading phase and throughout the study. Since this study is blinded, the research personnel will not know which supplement you are given and will therefore ensure everyone is following the same procedures.
  * Loading here means to consume more than the daily amount of supplement. This visit will have participants consume 5g twice in one day and twice more at home. This is a normal practice and standard use of the supplement.
  * If you are not in the control group, you will further be randomized into one of four possible supplementation groups. These groups will be double blinded and randomized into either placebo or creatine supplementation. Creatine monohydrate powder (Muscle Feast, Creapure®) will be used for the active supplement group. Dextrose powder (sugar) will be used for the placebo group.
  * The supplement and placebo are flavorless and odorless powder.
  Interventions: Other: Exercise

INTERVENTIONS:
Dietary Supplement: Creatine Monohydrate — Creatine supplementation for 8 weeks, 5g daily. A 5 day loading phase will be implemented with 20g daily for 5 days.
  Arms: Creatine and Blood Flow Restriction Exercise; Creatine and No-BFR with Training
Device: Blood Flow Restriction — Blood Flow Restriction Cuffs applied during exercise
  Arms: Creatine and Blood Flow Restriction Exercise; Placebo and Blood Flow Restriction Exercise
Other: Exercise — Participants will exercise
  Arms: Placebo and No-BFR with Training

SUMMARY:
This research is examining the changes in muscle size, muscle function, body composition, strength, and blood vessel health. Specifically, the changes in these variables over the course of 8 weeks of training with or without blood flow restriction (BFR) and the supplementation of creatine or placebo (dextrose, a sugar in the form of a powder which is the standard placebo). Creatine monohydrate (Cr) is the most popular supplement for athletes and benefits all populations, however women are still very hesitant to take it due to the misconception of weight gain. This study will look to measure those muscle and body changes with exercise.

DETAILED DESCRIPTION:
We expect that you will be in this research study for an estimated 10 weeks, with 27 visits total. You will be asked to complete questionnaires, blood draws, and perform exercises using exercise machines for testing the strength of your legs while using a blood pressure cuff during some of these exercises. Other tests in this study will measure hydration (water in your system) status, your nervous system, and body composition percentage (bone/muscle tissue/fat tissue). Specifically, you will be asked to attend:

* 1 consent visit with familiarization (60min)
* 1 baseline assessment with a blood sample (60min)
* 1 baseline strength assessment (45min)
* 2 creatine supplementation loading day visits (15min)
* 1 post loading assessment with a blood sample (60min)
* 1 post loading strength assessment (45min)
* 16 training days (60min each) two of which will have blood samples (+70min)
* 1-4wk follow up assessment (45min)
* 1 4wk follow up strength assessment (45min)
* 1 posttest assessment (45min)
* 1 posttest strength assessment (45min)

ELIGIBILITY:
Inclusion Criteria:

* Are female between the ages of 18 to 35
* Recreationally active, defined as meeting the ACSM standards for recreationally active individuals of participating in physical activity ≥ 150 minutes exercise/week.
* Not following a resistance training program
* Are Not currently taking creatine monohydrate or have not taken it in the last 6 weeks
* No known cardiovascular, pulmonary, metabolic, muscular, and/or coronary heart disease (i.e. heart failure, diabetes, COPD, etc.)
* Do not regularly use prescription medication (not including contraceptives)
* Are not currently seeking medical care.
* Are not currently pregnant.

Exclusion Criteria:

* Taking creatine or has taken creatine in the last 6 weeks
* Currently resistance training
* Pregnant

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Strength | Pre, 5-Days post loading, 4wk, 8wk
  isokinetic dynanometer
Body Composition | Pre, 5-Days post loading, 4wk, 8wk
  BIS, BodPod
Neuromuscular Function | Pre, 5-Days post loading, 4wk, 8wk
  EMG
Endothelial Function | Pre, 5-Days post loading, 4wk, 8wk
  Flow Mediated Dilation

SECONDARY OUTCOMES:
Mood States | Pre, 5-Days post loading, 4wk, 8wk
  Mood Assessed via administration of the POMS Questionnaire. 58 words or phrases are presented in a Likert format questionnaire reflecting how the subject feels at the time of completing the questionnaire. Scores range from 0 (Not at all) to 4 (Extremely). Tension, depression, anger, vigor, fatigue, confusion and total mood disturbance (TMD) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Paola M Rivera, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No